CLINICAL TRIAL: NCT05923931
Title: Non-inferiority Study of the Effect of Non-cooling Blanket on Body Temperature in Patients With Heat Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Yiwu Central Hospital (Other); Jinhua People's Hospital (Unknown); Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); Lanxi People's Hospital (Other); Hangzhou Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0508
Record Dates: First submitted 2023-05-23; First posted 2023-06-28 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Heat Stroke
Keywords: heat stroke, cooling blanket, cooling rate, outcomes
MeSH Terms: conditions — Heat Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-cooling blanket group (Experimental): Cooling body temperature by: control the temperature of the emergency room to 20-24℃, 4℃ fluid infusion, ice packs, evaporation, convection, etc.
  Interventions: Device: non-cooling blanket
- Cooling blanket group (Active Comparator): On the basis of the cooling methods of non-cooling blanket group, combine the cooling blanket to cool down. The cooling blanket is required to be activated within 30min after admission. The blanket temperature will be set at 4-10℃, and the target body temperature is 38℃.
  Interventions: Device: cooling blanket

INTERVENTIONS:
Device: cooling blanket — On the basis of the cooling methods of non-cooling blanket group, combine the cooling blanket to cool down. The cooling blanket is required to be activated within 30min after admission. The blanket temperature will be set at 4-10℃, and the target body temperature is 38℃.
  Arms: Cooling blanket group
Device: non-cooling blanket — Patients do not receive cooling blanket according to randomization. Cooling body temperature by: control the temperature of the emergency room to 20-24℃, 4℃ fluid infusion, ice packs, evaporation, convection,etc.
  Arms: non-cooling blanket group

SUMMARY:
The goal of this clinical trial is to test the cooling effect of cooling blanket in patients with heat stroke. The main questions it aims to answer are:

* the cooling rate of cooling blanket in patients with heat stroke
* the relationship between cooling blanket and outcomes in patients with heat stroke

Participants will accept the cooling blanket or non-cooling blanket according to the randomization group.

Researchers will compare cooling rate and outcomes to see if the cooling blanket can accelerate the cooling speed and improve the prognosis of patients in heat stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* diagnosed as heat stroke
* informed consent of patients or family members

Exclusion Criteria:

* need immediate cardiopulmonary resuscitation
* body temperature <39.5℃ on admission
* with the underlying disease of severe organ damage
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
cooling rate at 0.5 hours | 0.5 hours
  The cooling rate of 0.5h was calculated by the initial temperature and the 0.5 hours temperature.
Body temperature of 0.5 hours | 0.5 hours after admission to emergency department
  Body temperature of 0.5 hours referred to the temperature value obtained 5 min before and after 0.5 hour.

SECONDARY OUTCOMES:
Body temperature of 2 hours | 2 hours
  Body temperature of 2 hours referred to the temperature value obtained 20 min before and after 2 hours.
incidence of organ damage | up to 90 days
  number of participants with organ damage, including but not limited to brain, lung, heart, kidney, liver, and coagulation function
length of ICU stay | up to 90 days
  The length patient stay at ICU
in-hospital mortality | up to 90 days
  number of participants dead in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Lan Chen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - Yongkang First People's Hospital, Guli, Zhejiang
  - Yiwu Central Hospital, Yiwu, Zhejiang
  - Dongyang People's Hospital, Dongyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - Jinhua People's Hospital, Jinhua
  - Lanxi People's Hospital, Lanxi